CLINICAL TRIAL: NCT02050724
Title: Thorakoskopische Handheld-SPECT Gesteuerte Ektomie Von Radioaktiv-markierten Pulmonalen Rundherden. Proof of Feasibility of Thoracoscopic Ectomy of Radioactively Marked Pulmonary Nodules With the Help of Free-hand SPECT.
Brief Title: ThoHSpEkt Thoracoscopic Ectomy of Radioactively Marked Pulmonary Nodules With Free-hand SPECT
Acronym: ThoHSpEkt
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Ende of part 1. Only few patients in part 2 enrolled
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Joachim Müller, Head of Department, Cantonal Hospital of St. Gallen
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CTU 12/048
Record Dates: First submitted 2013-11-28; First posted 2014-01-31 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Solitary Pulmonary Nodule; Bronchial Neoplasms
Keywords: Solitary Pulmonary Nodule; Thoracoscopy; Thoracic Surgery; Video-Assisted; Radioactive Tracers; Radioguided surgery; Handheld-SPECT
MeSH Terms: conditions — Solitary Pulmonary Nodule; Bronchial Neoplasms | interventions — Technetium Tc 99m Aggregated Albumin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT guided labelling (Experimental): CT guided radioactive labelling of pulmonary nodules followed by handheld-SPECT guided thoracoscopic surgery.
  Interventions: Drug: Radioactive labelling of pulmonary nodules; Device: CT guided radioactive labelling
- Electromagnetic bronchoscopic labelling (Experimental): Electromagnetic guided bronchoscopic labeling of pulmonary nodules followed by handheld-SPECT guided thoracoscopic surgery.
  Interventions: Drug: Radioactive labelling of pulmonary nodules; Device: Electromagnetic guided bronchoscopic radioactive labelling

INTERVENTIONS:
Drug: Radioactive labelling of pulmonary nodules — Application directly into a pulmonary nodule
  Other Names: Tc-99m MAA (Maasol GE)
Device: CT guided radioactive labelling — CT guided puncture is a standard procedure in radiology. In this study it is used to mark pulmonary nodules for the following thoracoscopic surgery, done with a handheld-SPECT device.
  Other Names: CT GE (PET-CT Discovery)
  Arms: CT guided labelling
Device: Electromagnetic guided bronchoscopic radioactive labelling — Electromagnetic guided bronchoscopy is a standard procedure. In this study it is used to mark pulmonary nodules.
  Other Names: iLogic, Firme SuperDimension
  Arms: Electromagnetic bronchoscopic labelling

SUMMARY:
Title ThoHSpEkt

Study Design Pilot Study concerning the technical operative methods and a phase II study concerning the radiopharmaceutical (therapeutic-explorative study with an approved drug in a new indication)

Location Kantonsspital St.Gallen

Aim Proof of feasibility of thoracoscopic ectomy of radioactively marked pulmonary nodules with the help of free-hand SPECT.

Background In the Cantonal Hospital of St.Gallen an average of 30 - 40 patients will be operated with thoracoscopic ectomy for a pulmonary nodule. When localisation of the nodule is not possible a switch to minithoracotomy is performed.

Study intervention Marking of pulmonary nodules with radioactivity. Free-hand SPECT guided surgery

Risks Risks of bronchoscopic or CT-intervention Radiation risk (minimal)

Rational for patient number 10 patients for each group are enough to prove the feasibility, to manage difficulties and to record complications

Duration approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* Planed thoracoscopic surgery of a pulmonary nodule
* Informed consent

Exclusion Criteria:

* mental incapacity
* contraindications for this treatment
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Successful thoracoscopic ectomies | 1 week
  Rate of successful thoracoscopic ectomies (i.e. without reversion to (mini-)thoracotomy and without any complications)

SECONDARY OUTCOMES:
CT labelling | 1 day
  Success rate of CT labelling
CT Labelling complications | 1 day
  complication rate attributable to CT labelling
Successful labeling using electro-magnetically navigated bronchoscopy | 1 day
  Rate of successful labeling using electro-magnetically navigated bronchoscopy
Complications after labeling using electro-magnetically navigated bronchoscopy | 1 day
  Complication rate after labeling using electro-magnetically navigated bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Müller, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital St.Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Derived] Muller J, Putora PM, Schneider T, Zeisel C, Brutsche M, Baty F, Markus A, Kick J. Handheld single photon emission computed tomography (handheld SPECT) navigated video-assisted thoracoscopic surgery of computer tomography-guided radioactively marked pulmonary lesions. Interact Cardiovasc Thorac Surg. 2016 Sep;23(3):345-50. doi: 10.1093/icvts/ivw136. Epub 2016 May 20. PMID 27207315